CLINICAL TRIAL: NCT01003067
Title: Intraperitoneal Mesh-Implementation After Laparotomy to Reduce Risk of Incisional Hernia: a Prospective Randomized Controlled Trial
Brief Title: Intraperitoneal Mesh-Implementation After Laparotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Principal Investigator, Christoph A. Maurer, MD, Prof. Dr. med. Christoph A. Maurer, Kantonsspital Liestal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 364/07
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Mesh (No Intervention)
- Mesh Implementation (Experimental)
  Interventions: Device: Mesh implementation

INTERVENTIONS:
Device: Mesh implementation — Prophylactic intraperitoneal mesh implantation in laparoscopic surgery to prevent incisional hernia.
  Arms: Mesh Implementation

SUMMARY:
Aim of the study is to evaluate the risk reduction of intraperitoneal mesh-implementation after laparotomy (Group 1) in a randomized control trial compared with patients with standard abdominal closure (Everett-suture). This is the primary endpoint. Second endpoints are the feasibility of mesh-implementation even after colorectal surgery, find risk factors for wound infection and incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Median Laparotomy

Exclusion Criteria:

* Bowel perforation
* Pregnancy
* Palliative surgery
* Drug abuse
* Age under 18
* Mental disability
* Allergy to mesh components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2008-03; Primary Completion 2013-05 (Actual); Study Completion 2020-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Liestal, Liestal, Basel-Landschaft, Switzerland

REFERENCES:
- [Derived] Glauser PM, Brosi P, Speich B, Kaser SA, Heigl A, Rosenberg R, Maurer CA. Prophylactic Intraperitoneal Onlay Mesh Following Midline Laparotomy-Long-Term Results of a Randomized Controlled Trial. World J Surg. 2019 Jul;43(7):1669-1675. doi: 10.1007/s00268-019-04964-6. PMID 30824961
- [Derived] Brosi P, Glauser PM, Speich B, Kaser SA, Maurer CA. Prophylactic Intraperitoneal Onlay Mesh Reinforcement Reduces the Risk of Incisional Hernia, Two-Year Results of a Randomized Clinical Trial. World J Surg. 2018 Jun;42(6):1687-1694. doi: 10.1007/s00268-017-4363-2. PMID 29159603

RESULTS

PARTICIPANT FLOW:
Groups:
- No Mesh: conventional abdominal closure with a suture
Period: Overall Study
Arm/Group | No Mesh | Mesh Implementation
Started | 136 | 131
Completed | 103 | 107
Not Completed | 33 | 24

BASELINE CHARACTERISTICS:
Groups:
- No Mesh: The closure technique consisted of a single-layer continuous suture technique with picking up all layers of the abdominal wall apart from subcutaneous fat and skin (peritoneum, posterior rectus sheath, rectus muscle and anterior rectus sheath).
- Total: Total of all reporting groups
Arm/Group | No Mesh | Mesh Implementation | Total
Number analyzed (Participants) | 136 | 131 | 267
Age, Customized [Mean (Standard Deviation); unit: years] | 65.1 (2) | 64.1 (2.3) | 64.5 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 71 | 151
  Male | 56 | 60 | 116
Region of Enrollment [Number; unit: participants]
  Switzerland | 136 | 131 | 267

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incisional Hernia At 2 Years Following Median Laparotomy
Description: Primary endpoint was the incidence of incisional hernias at 2 years following midline laparotomy.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | No Mesh | Mesh Implementation
Number analyzed (Participants) | 103 | 107
participants | 40 | 18

2. Secondary Outcome: Feasibility of Mesh-implementation Even After Colorectal Surgery, Find Risk Factors for Wound Infection and Incisional Hernia.
Description: Secondary endpoints are the feasibility, the safety of the mesh stripe implantation including postoperative pain, and the incidence of incisional hernias at 5 years.
Time Frame: 5 Years
Reporting Status: Not Posted, anticipated posting 2020-06

ADVERSE EVENTS:
Arm/Group | No Mesh | Mesh Implementation
All-Cause Mortality (participants affected / at risk) | 10/136 | 4/131
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/131
Other Adverse Events (participants affected / at risk) | 0/136 | 2/131
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Mesh (N=136) | Mesh Implementation (N=131)
Bowel Fistulation (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes